CLINICAL TRIAL: NCT02709356
Title: Proof of Concepts: Can a Supplement Ketogenic Based MCT Oil Increases Cerebral Capture Ketones in People With Alzheimer's Disease?
Brief Title: Medium Chain Triglycerides and Brain Metabolism in Alzheimer's Disease
Acronym: MCT-MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fondation Vitae (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-547
Record Dates: First submitted 2016-02-01; First posted 2016-03-16 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2017-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alzheimer's disease (Experimental): Patients with mild Alzheimer's disease.
  1-month of 60-40 MCT oil and 1-month of C8 MCT oil (order of the two intervention are randomized)
  Interventions: Dietary Supplement: 1-month of 60-40 MCT oil; Dietary Supplement: 1-month of C8 MCT oil
- Controls (Experimental): Healthy elderly people
  1-month of 60-40 MCT oil and 1-month of C8 MCT oil (order of the two intervention are randomized)
  Interventions: Dietary Supplement: 1-month of 60-40 MCT oil; Dietary Supplement: 1-month of C8 MCT oil

INTERVENTIONS:
Dietary Supplement: 1-month of 60-40 MCT oil — 1-month supplementation of 30 g MCT oil (60% C10 + 40% C8)/day
Dietary Supplement: 1-month of C8 MCT oil — 1-month supplementation of 30 g MCT oil (100% C8)/day (1-month of C8 MCT oïl)

SUMMARY:
Evaluate and compare the changes in brain ketone and glucose uptake after taking two different MCT oil emulsions (60-40 oil or C8 oil) for one month, in a group of people with Alzheimer's disease and a control group.

DETAILED DESCRIPTION:
Based on a PET/MRI protocol, the aim of this study is to evaluate and compare the response to the dietary supplementation of two different MCT oils (60% C10 + 40% C8 or 100 % C8) in two groups, patients with Alzheimer's disease and healthy elderly people (N=10/group). After a baseline evaluation, participant will test one of the supplements during two successive periods of one month; each period of time ending with 18F-FDG and 11C-acetoacetate PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Good general health for Control group
* Diagnosis of Alzheimer's disease (NINCDS-ADRDA criteria) for AD group

Exclusion Criteria:

* Depression
* Medical or psychiatric conditions that could interfere with study participation
* Fasting plasma glucose ≥7.0 mM (diabetes or prediabetes)
* Already on MCT supplementation
* Clinically-significant gastrointestinal disease/conditions
* Clinically-significant liver disease/dysfunction
* Clinically-significant renal disease/dysfunction
* Clinically-significant cardiac disease/conditions
* Hypertension
* Uncontrolled dyslipidaemia
* Vitamin B12 deficiency
* Structured physical activity (more than 3 times/week)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Quantification of brain glucose uptake | 1-month
  Brain glucose uptake (umol/100g/min) using 18-FDG PET scan
Quantification of brain acetoacetate uptake | 1-month
  Brain acetoacetate uptake (umol/100g/min) using 11C-AcAc PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, PhD, Principal Investigator — Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS) - Université de Sherbrooke
Locations (1):
- Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided